CLINICAL TRIAL: NCT02160873
Title: Effect of Nighttime Feeding on Morning Performance in Female Endurance Athletes
Brief Title: Nighttime Feeding and Morning Endurance Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CHMK-1415
Record Dates: First submitted 2014-04-01; First posted 2014-06-11 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Poor Performance Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chocolate milk (Experimental): In this arm, subjects receive chocolate milk
  Interventions: Other: chocolate milk
- flavor-matched placebo (Placebo Comparator): In this arm, subjects receive a flavor-matched placebo
  Interventions: Other: flavor-matched placebo

INTERVENTIONS:
Other: chocolate milk — 12 oz, 7-8 hours prior to exercise trial (night before)
  Arms: chocolate milk
Other: flavor-matched placebo — 12 oz, non-caloric flavor-matched placebo
  Arms: flavor-matched placebo

SUMMARY:
The purpose of this study is to investigate the influence of a nighttime feeding on next morning running performance, hydration status, and exercise metabolism in female endurance athletes. Specifically, the effect of a chocolate milk beverage will be examined versus a non-nutritive, flavor-matched placebo. The investigators hypothesize that the nighttime consumption of chocolate milk, a whole food complex, will result in improved next morning running performance versus placebo. Secondarily, the investigators hypothesize that any potential positive performance outcomes from the chocolate milk treatment may be due to an enhanced pre-exercise hydration status or improved exercise metabolism.

DETAILED DESCRIPTION:
This study will be interventional in nature and employ a crossover, randomized, double-blinded approach. This study will include a maximal oxygen uptake test and three trials: one familiarization trial, and two experimental trials. The familiarization will serve as a practice test to minimize any training effects between experimental trials. The experimental trials will be completed within a 2-week period determined by the luteal phase of the menstrual cycle (days 15-28 of the menstrual cycle, with day 1 being the first day of menstruation). A minimum of 48-72 hours will be provided between testing days.

Experimental trials will consist of baseline testing (height, weight, urinalysis, resting metabolic rate), followed by a treadmill performance protocol. Participants will complete a 3-stage incremental exercise test (at 55%, 65%, and 75% of maximal oxygen uptake respectively). Metabolic data will be collected during this time. Participants will then complete a 10-kilometer running time trial in which markers of intensity are monitored at various time points (blood glucose, blood lactate, heart rate, rating of perceived exertion). Participants and primary researchers will be blinded to all time and speed data. Distance will be the only known measure of progress. Additional blood, urine, and body weight measures will be taken immediately post exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 18 and 40 years old
* Consistently use oral contraceptives (greater than 2 months) or be considered eumenorrheic without oral contraceptive use
* 'Moderately trained,' defined as a weekly mileage ≥ 25 miles for at least 6 months, and a VO2max ≥ 45 ml/kg/min

Exclusion Criteria:

* Lactose intolerant
* Smokers
* Uncontrolled thyroid conditions
* Uses anti-inflammatory drugs or any dietary supplements intended to improve performance
* Have musculoskeletal injury that could limit performance

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ormsbee, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects were recruited from the Tallahassee running community.
Pre-assignment Details: Subjects were randomized to receive either chocolate milk first or placebo first. In between exercise trials, there was a 7-day washout period.
Groups:
- Chocolate Milk, Then Placebo: Subjects received chocolate milk: 12 oz, 7-8 hours prior to exercise trial (night before). Thereafter, there was a 7 day washout period. Then, subjects received the placebo beverage 7-8 hours prior to the exercise trial.
- Flavor-matched Placebo, Then Chocolate Milk.: Subjects received flavor-matched placebo: 12 oz, 7-8 hours prior to exercise trial (night before). Thereafter, there was a 7 day washout period. Then, subjects received 12 oz of chocolate milk 7-8 hours prior to exercise.
Period: Overall Study
Arm/Group | Chocolate Milk, Then Placebo | Flavor-matched Placebo, Then Chocolate Milk.
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Trained runners and triathletes
Groups:
- Chocolate Milk First, Then Placebo: chocolate milk: 12 oz, 7-8 hours prior to exercise trial (night before) followed by a 7-day washout, then placebo 7-8 hours prior to exercise trial.
- Flavor-matched Placebo, Then Chocolate Milk: flavor-matched placebo: 12 oz, 7-8 hours prior to exercise trial (night before) followed by a 7-day washout, then chocolate milk 7-8 hours prior to exercise trial.
- Total: Total of all reporting groups
Arm/Group | Chocolate Milk First, Then Placebo | Flavor-matched Placebo, Then Chocolate Milk | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (6.4) | 29.3 (7.1) | 29.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Body fat (%) [Mean (Standard Deviation); unit: %] | 21.4 (5.7) | 22.1 (5.0) | 21.8 (5.1)
Maximal oxygen consumption (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] | 51.8 (4.1) | 53.8 (4.5) | 52.8 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Running Performance
Description: 10K time trial on a treadmill
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Flavor-matched Placebo: flavor-matched placebo: 12 oz, 7-8 hours prior to exercise trial (night before)
Arm/Group | Chocolate Milk | Flavor-matched Placebo
Number analyzed (Participants) | 12 | 12
minutes | 52.8 (8.0) | 52.8 (8.4)

2. Secondary Outcome: Urine Specific Gravity
Description: Changes in urine specific gravity will be measured pre and post a 10K time trial run on a treadmill
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Urine specific gravity
Groups:
- Chocolate Milk: In this arm, subjects receive chocolate milk (in a cross-over design)
  chocolate milk: 12 oz, 7-8 hours prior to exercise trial (night before)
- Flavor-matched Placebo: In this arm, subjects receive a flavor-matched placebo (in a cross-over design)
  flavor-matched placebo: 12 oz, non-caloric flavor-matched placebo
Arm/Group | Chocolate Milk | Flavor-matched Placebo
Number analyzed (Participants) | 12 | 12
Urine specific gravity | -0.005 (0.008) | -0.002 (0.009)

3. Other Pre Specified Outcome: Exercise Metabolism
Description: Indirect calorimetry will be used to assess macronutrient use during exercise via the respiratory exchange ratio
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Respiratory exchange ratio
Arm/Group | Chocolate Milk | Flavor-matched Placebo
Number analyzed (Participants) | 12 | 12
Respiratory exchange ratio
  55% VO2max | 0.84 (0.04) | 0.82 (0.04)
  65% VO2max | 0.85 (0.04) | 0.83 (0.03)
  75% VO2max | 0.87 (0.03) | 0.85 (0.03)

4. Secondary Outcome: Urine Volume
Description: Measurement of total urine output.
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: mililiters
Groups:
- Chocolate Milk: Subjects received chocolate milk: 12 oz, 7-8 hours prior to exercise trial (night before). Thereafter, there was a 7 day washout period. Then, subjects received the placebo beverage 7-8 hours prior to the exercise trial.
- Flavor-matched Placebo: Subjects received flavor-matched placebo: 12 oz, 7-8 hours prior to exercise trial (night before). Thereafter, there was a 7 day washout period. Then, subjects received 12 oz of chocolate milk 7-8 hours prior to exercise.
Arm/Group | Chocolate Milk | Flavor-matched Placebo
Number analyzed (Participants) | 12 | 12
mililiters | 718.07 (260.82) | 874.82 (179.6)

ADVERSE EVENTS:
Time Frame: Data was collected for 4 weeks.
Arm/Group | Chocolate Milk | Flavor-matched Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chocolate Milk (N=12) | Flavor-matched Placebo (N=12)
Reduced sleep quality (General disorders) | 4 (4) | 0 (0) — Subjects reported altered sleep quality and/or duration following intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No